CLINICAL TRIAL: NCT05971277
Title: Proof of Concept (POC) Prospective Observational Study to Test a Framework for Integration of Data Streams, Including Molecular Genomic Markers and Wearable Device Data in Patients Receiving Chemotherapy for Advanced Cancer
Brief Title: Home And Locally Observed - Tracking (HALO-Trak)
Acronym: HALO-Trak
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 150745; 312296 (Other: IRAS)
Record Dates: First submitted 2023-01-09; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-01

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genomic and microbiome analysis, statistical analysis
Oversight: FDA-regulated Drug: No

INTERVENTIONS:
Device: Halo Wearable data device — A wrist-worn tracker with heart-rate monitor and pedometer (step counter), as well as a mobile app.

SUMMARY:
The goal of this observational study is to collect biometric, HRQoL, immune response and genomic data continuously and intermittently during and after chemo or immunotherapy for the generation of a complex dataset using a platform which can aggregate different types of data collected over a time period and, to test the potential for analysis within and across data sets with linkage to clinical outcomes. The framework will have capabilities to integrate data from electronic medical records (EMRs) such as Epic, as well as digital streams including sensor, genomic, imaging and pathology. Such a platform can realise the potential for machine learning (ML) methodologies to address important cancer outcomes.

DETAILED DESCRIPTION:
The Investigators overarching aim is to determine the relationship between measures of physical performance status including heart rate and steps, health related quality of life (HRQoL) and genomic and immunogenomic phenotype on cancer outcomes in patients receiving chemotherapy or immunotherapy for haematological or metastatic cancer including renal (papillary, and RCC), breast, prostate, and other solid tumours. The primary objective is to test the feasibility of integrating diverse data streams (genomic, HR QoL and biometric) on a novel platform, capable of integrating data streams thus generating complex datasets for analyses using machine learning methodologies.

Secondary objectives will be to conduct exploratory analysis assessing the relationship between individual and combined data types and cancer outcomes.

Analysis using existing and novel computational models will be applied to the data to events in the acute and chronic setting that are common in patients diagnosed with cancer undergoing systemic therapy such as chemotherapy and immunotherapy. The outputs from this study will help inform future studies and trials designed to inform patients about their health status during cancer therapy

ELIGIBILITY:
Inclusion Criteria:

* ● A diagnosis of a metastatic or haematological cancer undergoing systemic therapy

  * Undergoing at least 1 planned cycle of chemotherapy or immunotherapy, according to standard of care practices.
  * Ability to understand and the willingness to sign a written informed consent.
  * Able to ambulate without assistance or walking aid.
  * Have an Android or iOS phone and willing to download the Ethera app

Exclusion Criteria:

* ● Physical disabilities that preclude daily walking

  * Inability to provide informed consent.
  * Unable to use and operate the Ethera Health Monitoring Smartphone App. (Apple or Android)
  * Medical or psychiatric condition which in the investigator's opinion would affect the successful completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will be receiving standard of care therapies and will be recruited from Oncology clinics once a diagnosis of metastatic or haematological cancers has been established and patients meet all the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | one month to 52 weeks
  To measure feasibility of data collection longitudinally in a patient cohort undergoing systemic therapy for metastatic or haematological cancer.
Remote monitoring data | one month to 52 weeks
  To collect activity (steps) and heart rate data. This will be collected using the Ethera Wellness app which participants will download onto their smartphone devices.
Biological sample data. This will include blood samples (30mls) maximum frequency will be monthly | one month to 52 weeks
  This will include blood samples (30mls) and stool samples maximum frequency will be monthly
Clinical Outcome data | one month to 52 weeks
  Data will be collected via an electronic case report form-
Quality of life Questionnaire | one month to 52 weeks
  EORTC QLQ C30- questionnaire will be collected monthly

CONTACTS AND LOCATIONS:
Locations (1):
- UCL London, London, United Kingdom